CLINICAL TRIAL: NCT02715180
Title: Optimum Hand Position During Cardiopulmonary Resuscitation: Comparing Expiration and Inspiration View of the Scout Film of the Low Dose Chest Computed Tomography
Brief Title: Optimum Hand Position During Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyuksool Kwon, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hear_position_01
Record Dates: First submitted 2016-03-14; First posted 2016-03-22 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Cardiopulmonary Resuscitation; Hand Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chest computed tomography (Other): Low dose chest computed tomography during expiration and inspiration
  Interventions: Radiation: low dose chest computed tomography

INTERVENTIONS:
Radiation: low dose chest computed tomography — All participants were evaluated 2 scout films during LDCT screenings. The first scout film was obtained while a participant was holding a comfortable expiration with the arms at down position, and the second scout film was obtained while a full inspiration with the arms at raised position. The axial images of LDCT were taken during participants' full inspiration. The radio-opaque marker was attached to the participants' skin where the lowest part of sternum was palpable, because the sternum moves according to the position of arms and respiration.

SUMMARY:
The almost evidences of the optimal hand position during compression had been based on chest computed tomography (CT) or chest plain films of patients for investigating the effective location for compressing the left ventricle of the heart during cardiopulmonary resuscitation (CPR).

However every study was conducted at full inspired state of respiration. A prospective cohort study to evaluate the proper hand position during CPR based on expired respiratory state CT as the health screening would be needed.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* no history of heart or lung disease
* no history of chest or abdominal surgery

Exclusion Criteria:

* abnormal findings in LDCT, which might influence inspiration or expiration, were excluded after image interpretation by the board certified radiologists

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
proper hand position during CPR using the scout film of low dose chest computed tomography | five months
  proper hand position during CPR based on comparison between expiration with the arms at down position and inspiration the arms at raised position.
  Measurement will be assessed with a length of xiphoid process to arbitrary center of heart

SECONDARY OUTCOMES:
predicted compressed organs in CPR using the scout film of low dose chest computed tomography Measurement will be assessed with scout film silhouette of organs under quarterly divided sternum. | five months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klouche K, Weil MH, Sun S, Tang W, Povoas H, Bisera J. Stroke volumes generated by precordial compression during cardiac resuscitation. Crit Care Med. 2002 Dec;30(12):2626-31. doi: 10.1097/00003246-200212000-00002. PMID 12483049
- [Background] Perkins GD, Handley AJ, Koster RW, Castren M, Smyth MA, Olasveengen T, Monsieurs KG, Raffay V, Grasner JT, Wenzel V, Ristagno G, Soar J; Adult basic life support and automated external defibrillation section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 2. Adult basic life support and automated external defibrillation. Resuscitation. 2015 Oct;95:81-99. doi: 10.1016/j.resuscitation.2015.07.015. Epub 2015 Oct 15. No abstract available. PMID 26477420
- [Background] Travers AH, Perkins GD, Berg RA, Castren M, Considine J, Escalante R, Gazmuri RJ, Koster RW, Lim SH, Nation KJ, Olasveengen TM, Sakamoto T, Sayre MR, Sierra A, Smyth MA, Stanton D, Vaillancourt C; Basic Life Support Chapter Collaborators. Part 3: Adult Basic Life Support and Automated External Defibrillation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S51-83. doi: 10.1161/CIR.0000000000000272. PMID 26472859
- [Background] Cha KC, Kim HJ, Shin HJ, Kim H, Lee KH, Hwang SO. Hemodynamic effect of external chest compressions at the lower end of the sternum in cardiac arrest patients. J Emerg Med. 2013 Mar;44(3):691-7. doi: 10.1016/j.jemermed.2012.09.026. Epub 2012 Dec 4. PMID 23218197
- [Background] Qvigstad E, Kramer-Johansen J, Tomte O, Skalhegg T, Sorensen O, Sunde K, Olasveengen TM. Clinical pilot study of different hand positions during manual chest compressions monitored with capnography. Resuscitation. 2013 Sep;84(9):1203-7. doi: 10.1016/j.resuscitation.2013.03.010. Epub 2013 Mar 15. PMID 23499897
- [Background] Orlowski JP. Optimum position for external cardiac compression in infants and young children. Ann Emerg Med. 1986 Jun;15(6):667-73. doi: 10.1016/s0196-0644(86)80423-1. PMID 3706857
- [Background] Pickard A, Darby M, Soar J. Radiological assessment of the adult chest: implications for chest compressions. Resuscitation. 2006 Dec;71(3):387-90. doi: 10.1016/j.resuscitation.2006.04.012. Epub 2006 Sep 18. PMID 16982125